CLINICAL TRIAL: NCT06222554
Title: Pilot/Feasibility Study Examining the Use of a Novel Immersive Motion Tracking Upper Extremity Exercise Program for Acute Hospitalized Patients
Brief Title: Examining the Use of a Novel Immersive Motion Tracking Upper Extremity Exercise Program for Acute Hospitalized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 23-01384
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Kidney Transplant; Liver Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients Hospitalized following Kidney or Liver Transplant (Experimental): Patients in the study will be introduced to the exercise software program and provided with a demonstration. Measurements will be taken at baseline (post-operation) and at the final study visit. Participants will remain in the study until the end of their hospital stay, typically no longer than 6 months post-operation.
  Interventions: Device: MoveMend Health

INTERVENTIONS:
Device: MoveMend Health — Software-based therapeutic tool that offers gamified exercises and activities. The device is designed for deployment on tablets. The core purpose of the device is to augment patient engagement and participation in their own rehabilitation by providing additional therapeutic interventions between formal occupational therapy sessions.

SUMMARY:
The objective of this study is to evaluate the feasibility of the MoveMend Health software program as an integrated supplement to traditional acute care/in-hospital occupational therapy for patients following liver and kidney transplants, as determined by recruitment rates, program completion, intervention adherence, safety incidence, and patient feedback on device/program performance.

ELIGIBILITY:
Inclusion Criteria:

* English speaking (software program is currently only available in English)
* Status post kidney or liver transplant this admission
* Physician orders for occupational therapy evaluation and treatment
* Orientation Log > 25
* Negative for delirium per the Confusion Assessment Method

Exclusion Criteria:

* Orthopedic or surgical precautions that limits shoulder range of motion beyond 90 degrees
* Upper extremity hemiplegia with inability to lift upper extremity against gravity
* Accommodation code of Intensive Care Unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Up to Month 6 Post-Operation
  Calculated by dividing the number of participants enrolled by the total number of patients contacted or screened.
Percentage of Participants who Complete Exercise Program | Up to Month 6 Post-Operation
  Percentage of enrolled participants who complete the interventional program.
Percentage of Participants who Adhere to Intervention | Up to Month 6 Post-Operation
  Measured by session duration and frequency, as recorded by the device. Participants will be classified as "adhering" or "not adhering."
Number of Adverse Events | Up to Month 6 Post-Operation
  Measured using data from participant's electronic medical record.

SECONDARY OUTCOMES:
Change in Activity Measure for Post-Acute Care (AMPAC) Score | Baseline, End of Hospital Stay (typically no more than 6 months post-operation)
  12-item assessment of basic mobility of inpatients. Each item is rated on a Likert scale from 1-4. The raw score is the sum of responses, which is converted to a T-score. The total score is a T-score ranging from 0 to 100; higher scores indicate greater mobility.
Change in Grip Strength | Baseline, End of Hospital Stay (typically no more than 6 months post-operation)
  Measured as the percentage change in grip strength between the baseline assessment and the final assessment at discharge.
Upper Extremity Range of Motion (ROM) Change | Baseline, End of Hospital Stay (typically no more than 6 months post-operation)
  Measured as the change in degrees of ROM at the shoulder and elbow as measured by a goniometer from baseline to discharge.
Change in EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire Index Score | Baseline, End of Hospital Stay (typically no more than 6 months post-operation)
  The EQ-5D-5L is a self-reported health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. There are two components to the EQ-5D-5L: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a visual analogue scale (VAS) that measures health state. Overall scores range from 0 to 1, with low scores representing a higher level of dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: John Corcoran, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Gabrielle Berne, Gabrielle.berne@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Gabrielle.berne@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.